CLINICAL TRIAL: NCT05932771
Title: The Dose-response of Vitamin C-enriched Collagen on Markers of Collagen Synthesis in Healthy Young and Older Men and Women Following Resistance Exercise
Brief Title: Resistance Exercise and Hydrolyzed Collagen Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rob Erskine (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor-Investigator, Rob Erskine, Reader in Neuromuscular Physiology, Liverpool John Moores University
Organization: Liverpool John Moores University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18/SPS/059
Record Dates: First submitted 2023-05-26; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Diet, Food, and Nutrition
Keywords: Hydolyzed collagen; Resistance exercise; Collagen synthesis; Proline; Glycine

STUDY DESIGN:
Intervention Model Description: A double-blind, randomised cross-over design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Before commencing each experimental trial, a laboratory technician (independent to the study) made up the three doses of hydrolyzed collagen (HC) and randomly assigned the order of HC dose (Excel 2016, Microsoft, Washington, USA) for each participant. Also, for each trial, the technician recorded the date, randomly allocated trial number (1, 2 or 3) and corresponding HC dose to blind the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1.Trial for young male participants: Consuming hydrolyzed collagen (HC) with reistance exercise (Experimental): Young male participants consumed one of three different HC doses (0 grams, 15 grams, or 30 grams) with 4 sets of 10 repetitions of barbell back squat exercise at 10-repetition maximum load in a random order and a seven-day wash-out period interspersed between each trial.
  Interventions: Dietary Supplement: Experimental: Consumption of three different doses of hydrolyzed collagen (HC) with reistance exercise
- 2.Trial for young female participant: Consuming hydrolyzed collagen (HC) with reistance exercise (Experimental): The intervention procedure is exactly same as Arm 1 except for the number of visits. Young female participant was asked to visit the laboratory on four occasions during two consecutive months. Therefore, there were two trials in each month, where female participants' estrogen level was lower (i.e., onset of menses) or higher (i.e., ovulation). Dates for the trials were determined based on self-report of onset of menses and previous menstrual cycle length.
  Interventions: Dietary Supplement: Experimental: Consumption of two different doses of hydrolyzed collagen (HC) with reistance exercise
- 3.Trial for older male participants: Consuming hydrolyzed collagen (HC) with reistance exercise (Experimental): The age range of older male participants was 40 - 65 years. The intervention procedure is exactly same as Arm 1
  Interventions: Dietary Supplement: Experimental: Consumption of three different doses of hydrolyzed collagen (HC) with reistance exercise
- 4.Trial for older female participants: Consuming hydrolyzed collagen (HC) with reistance exercise (Experimental): The age range of older female participants was 40 - 65 years. The intervention procedure is exactly same as Arm 2
  Interventions: Dietary Supplement: Experimental: Consumption of two different doses of hydrolyzed collagen (HC) with reistance exercise

INTERVENTIONS:
Dietary Supplement: Experimental: Consumption of three different doses of hydrolyzed collagen (HC) with reistance exercise — Each trial lasts for seven hours and while participants consumed HC, performed resistance exercise and rested, 10 x 5 mL blood samples were collected from a superficial forearm vein using a cannula.
  All trials were performed at the same time of day (08:00 - 15:00).
  Different doses of HC (0 grams, 15 grams and 30 grams) and 50 milligrams vitamin C were dissolved with 250 milliliter water in an opaque bottle. To match calories of 30 grams HC, 34.1 grams and 15.4 grams maltodextrin was used in 0 grams HC and 15 grams HC respectively. Also to mask any potential difference in HC doses, 4 grams non-caloric sweetener was used in all HC doses.
  The details of nutritoinal supplements used are as follows:
  Hydrolysed collagen (Myprotein, Cheshire, UK), Vitamin C powder (Holland and Barrett Retail Limited, Warwickshire, UK), Maltodextrin (Myprotein, Cheshire, UK), and Non-caloric sweetener (Truvia®, SilverSpoon, London, UK)
  Other Names: Resistance exercise and collagen dose-response for male participants
  Arms: 1.Trial for young male participants: Consuming hydrolyzed collagen (HC) with reistance exercise; 3.Trial for older male participants: Consuming hydrolyzed collagen (HC) with reistance exercise
Dietary Supplement: Experimental: Consumption of two different doses of hydrolyzed collagen (HC) with reistance exercise — Each trial lasts for seven hours and while participants consumed HC, performed resistance exercise and rested, 10 x 5 mL blood samples were collected from a superficial forearm vein using a cannula.
  All trials were performed at the same time of day (08:00 - 15:00).
  Different doses of HC (0 grams and 30 grams) and 50 milligrams vitamin C were dissolved with 250 milliliter water in an opaque bottle. To match calories of 30 grams HC, 34.1 grams maltodextrin was used in 0 grams HC. Also to mask any potential difference in HC doses, 4 grams non-caloric sweetener was used in all HC doses.
  The details of nutritoinal supplements used are as follows:
  Hydrolysed collagen (Myprotein, Cheshire, UK), Vitamin C powder (Holland and Barrett Retail Limited, Warwickshire, UK), Maltodextrin (Myprotein, Cheshire, UK), and Non-caloric sweetener (Truvia®, SilverSpoon, London, UK)
  Other Names: Resistance exercise and collagen dose-response for female participants
  Arms: 2.Trial for young female participant: Consuming hydrolyzed collagen (HC) with reistance exercise; 4.Trial for older female participants: Consuming hydrolyzed collagen (HC) with reistance exercise

SUMMARY:
This study aimed to investigate the effect of different doses of hydrolyzed collagen (HC) with resistance exercise (RE) on whole body collagen synthesis in healthy young and older males and females.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of different doses of hydrolyzed collagen (HC) with resistance exercise (RE) on whole body collagen synthesis in healthy young and older males and females.

Healthy young and older males and females ingested 0 grams, 15 grams or 30 grams HC with 50 milligrams vitamin C 1h prior to performing four sets' barbell back-squat RE at 10-repetition maximum load, after which they rested for six hours. Blood samples were collected throughout each trial to analyse procollagen type Ⅰ N-terminal propeptide (PⅠNP, a biomarker of collagen synthesis) and β-isomerized C-terminal telopeptide of type I collagen (β-CTX, a biomarker of collagen breakdown) concentration, and the concentration of 18 amino acids that constitute collagen.

This is the first study to investigate the combined effect of different doses HC with high-intensity RE on whole body collagen synthesis in healthy young and older men and women. If 30 grams HC intake with RE does augment collagen synthesis more than RE alone, this suggests that long-term HC intake with chronic RE would be beneficial for tendon health, because collagen is the most abundant protein in tendon.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 months experienced in resistance exercise (regular back squat experience)
* Free from musculoskeletal injury
* Nullipara (a woman who has never given birth) (only for young female participatns)

Exclusion Criteria:

* Having a history of patellar tendon pathology
* Vegan
* Consumed nutritional supplements or medication purported to have beneficial effects on muscle-tendon properties (e.g. antioxidants, protein, etc.)
* Had a sustained a lower limb injury in the previous six months
* Smoker/vaper
* <18 or >40 years old (only for young participants)
* <40 ro >65 years old (only for older participants)
* Having an irregular menstrual cycle (only for young female participants)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in a marker of collagen synthesis | at rest immediately prior to HC ingestion, 0.5-hour post RE, 1-hour post RE, 2-hour post RE, 4-hour post RE and 6-hour post RE
  Serum procollagen type Ⅰ N-terminal propeptide (PⅠNP) concentrations were measured following 0 grams, 15 grams or 30 grams hydrolyzed collagen (HC) intake with resistnace exercise (RE) during all trials.
Change in a marker of collagen breakdown | at rest immediately prior to HC ingestion and 6-hour post RE
  Plasma β-isomerized C-terminal telopeptide of type I collagen (β-CTX) concentrations were measured following 0 grams, 15 grams or 30 grams hydrolyzed collagen (HC) intake with resistnace exercise (RE) during all trials.
Changes in amino acids concentrations in blood | at rest immediately prior to HC ingestion, 0.5-hour post HC ingestion, 1-hour post HC ingestion, 0.5-hour post RE, 1-hour post RE, 2-hour post RE, 4-hour post RE and 6-hour post RE
  Concentration of serum amino acids that constitute collagen was measured following 0 grams, 15 grams or 30 grams hydrolyzed collagen (HC) intake with resistnace exercise (RE) during all trials.

SECONDARY OUTCOMES:
Estrogen concentrations in women in each trial | at rest immediately prior to HC ingestion
  Concentrations of estrogen (17β-estradiol) was measured in each trial.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Erskine, PhD, Study Director — Liverpool John Moores University; Joonsung Lee, MSc, Principal Investigator — Liverpool John Moores University; Christopher Nulty, Principal Investigator — Liverpool John Moores University
Locations (1):
- Dr Rob Erskine, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT05932771/Prot_SAP_ICF_000.pdf